CLINICAL TRIAL: NCT06575257
Title: Neoadjuvant ADT +/- Darolutamide Followed by Radical Prostatectomy for High-risk Prostate Cancer: a Randomized, Open Label Trial
Brief Title: Neoadjuvant Therapy of Darolutamide Plus ADT for High Risk Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242118-C-1
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Darolutamide Plus ADT (Experimental): All participants in this arm will receive luteinizing hormone releasing hormone analogue (LHRHa) plus Darolutamide. Goserelin 3.6 mg will be used once per 4 weeks. Darolutamide will be administered orally as 600 mg twice a day. Subjects will continue to take Darolutamide Plus Goserelin for 12 weeks before radical prostatectomy
  Interventions: Drug: Darolutamide; Drug: Goserelin 3.6 mg
- ADT alone (Experimental): All participants in this arm will receive LHRHa alone for 12 weeks before receiving radical prostatectomy. Goserelin 3.6 mg will be administered once per 4 weeks.
  Interventions: Drug: Goserelin 3.6 mg

INTERVENTIONS:
Drug: Darolutamide — 600 mg orally twice daily for 12 weeks before radical prostatectomy
  Arms: Darolutamide Plus ADT
Drug: Goserelin 3.6 mg — 3.6 mg goserelin hypodermic once per 4 weeks

SUMMARY:
The purpose of this study is to determine if treatment with Darolutamide plus androgen deprivation therapy (ADT) before radical prostatectomy (RP) with pelvic lymph node dissection (pLND) in participants with high-risk localized or locally advanced prostate cancer results in an improvement in pathological complete response (pCR) rate and pathological tumor volume with minimal residual disease (MRD)) as compared to ADT.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 and ≤75 years of age.
* All patients must have a histologically or cytologically diagnosis of prostate cancer and must be eligible for radical prostatectomy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score ≤1.
* All patients must complete mpMRI or 68Ga-PSMA PET / CT before and after neoadjuvant treatment.
* All patients must undergo thorough tumor staging and meet one of the following criteria: 1. multi-parameter MRI or PSMA PET / CT shows clinical staging of primary tumor ≥ cT2c or cN+or locally advanced, 2. Gleason score of primary tumor ≥ 8, 3. prostate specific antigen (PSA) ≥20 ng/ml.
* Patients must have adequate organ function as defined by the following criteria(within 28 days prior to registration):

white blood cell (WBC) ≥ 4.0 × 109 / L platelets≥ 100 × 109 / L hemoglobin ≥ 9 g / dL international normalized ratio (INR) < 1.5. total bilirubin (TBIL)≤1.5 x upper limit of normal (ULN) SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN serum creatinine ≤2×ULN

* Patients must participate voluntarily and sign an informed consent form (ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.

Exclusion Criteria:

* clinical or radiological evidence of regional or extra-regional lymph node metastases or bone metastases or visceral metastases.
* Prior androgen deprivation therapy (medical or surgical) or focal treatment of prostate cancer or prostate cancer radiotherapy or prostate cancer chemotherapy.
* severe or uncontrolled concurrent infections.
* New York Heart Association Class III or IV congestive heart failure at the time of screening.
* uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
* Patients with mental illness, mental disability or inability to give informed consent are not eligible.
* Patients have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | After 12 weeks of neoadjuvant therapy + RP + PLND
  The proportion of subjects with no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy
Proportion of Subjects With Minimal Residual Disease | After 12 weeks of neoadjuvant therapy + RP + PLND
  The proportion of subjects that have residual tumors with maximum diameter of 5 mm or less after radical prostatectomy

SECONDARY OUTCOMES:
Rate of Stage Degradation | After 12 weeks of neoadjuvant therapy + RP + PLND
  Clinical or pathological stage degradation after neoadjuvant therapy
Rate of Positive Surgical Margins | After 12 weeks of neoadjuvant therapy + RP + PLND
  The proportion of subjects with positive surgical margins after radical prostatectomy
Rate of Complete Serum Remission | After 12 weeks of neoadjuvant therapy
  The proportion of subjects whose PSA is less than or equal to 0.2 ng/ml after 3 months of treatment
Proportion of subjects without PSA progression | 2 years after RP
  The proportion of subjects whose PSA has never gone below 1 ng/ml or who receive any radiotherapy or systemic treatment after radical prostatectomy
Imaging Response Rate | After 12 weeks of neoadjuvant therapy
  The proportion of subjects whose primary tumor is in complete remission on imaging or residual tumor's maximum diameter is less than 0.5cm
Recovery time of urinary continence (day) | 1 years after RP
  The recovery time of urinary continence (day) after radical prostatectomy, defined as 0 pad/day.
biochemical recurrence-free survival (bRFS) | 3 years after RP
  biochemical recurrence-free survival (bRFS) defined as time to PSA ≥ 0.2 ng/ml after radical prostatectomy.
metastasis-free survival (MFS) | 5 years after RP
  time from date of randomization to date of evidence of systemic disease on bone scan or cross-sectional imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Qin, MD, Principal Investigator — The First Affillated Hospital, the Air Force Medical University
Locations (1):
- The First Affillated Hospital, the Air Force Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No